CLINICAL TRIAL: NCT01544400
Title: Description and Evaluation of Eating Disorders in Elite Athletes
Brief Title: Description and Evaluation of Eating Disorders in Elite Athletes (TCA SHN)
Acronym: TCA SHN
Status: Terminated | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/09/03-V
Record Dates: First submitted 2012-02-17; First posted 2012-03-05 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Eating Disorders; Anorexia Nervosa; Boulimia Nervosa; Binge Eating Disorders
Keywords: reverse anorexia,; anorexia athletics
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Athletes in particular elite athletes have obsessional food and body concerns, in bond with a worship of the performance more and more invading, which lead to clinical and subclinical eating disorders. These eating disorders differ according to the disciplines and are difficult to diagnose in athletes because there are insufficiently described.

Our aim at estimating the frequency of eating disorders in athletes and describing eating disorders by means of somatic, dietetic and psychological evaluations.

ELIGIBILITY:
Inclusion Criteria:

* to have at least 12 years
* to be registered on the high level sportsmen list or to be in access to high level sport
* to have obtained the non opposition of the athlete if he is major (if not the legal person in charge of the athlete have to give is non opposition).
* to be affiliated to social security

Exclusion Criteria:

* presenting obvious cognitive disturbance
* not able to understand or/ and to read French language
* pregnant women
* subject under tutelage

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Athletes registered on the high level sportsmen list or in access to high level sport
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Presence of eating disorder | 1 day
  A subject presents an eating disorder if at least one of the tree clinical investigators (somatician, dietician, psychologist) mark it.
  Eating disorders will be described by:
  Dietetic consultation, Somatic examination, Psychological evaluation

SECONDARY OUTCOMES:
Presence of eating disorder according to the psychologist, dietician and the somatician | 1 day
  Presence of eating disorder according to the psychologist, dietician and the somatician
Sociodemographic variables | 1 day
  age, sex, sporting discipline exercised
Doping conduits variables | 1 day
  age of onset of consumption (PAP support products performance) legal and illegal, current frequency of consumption of PAP licit and illicit consumption as problematic or not the patient.
Investment in practice sporting variables | 1 day
  Desired level of sports, number of hours per week over the last 4 weeks, up / concern of the sport.
Addictives and psychiatric comorbidity | 1 day
  anxiety disorders, depression and sleep disorders Scale : GEEMS, EDI, EDS-R

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Pretagut, Principal Investigator — Nantes University Hospital; Serge Lise, Principal Investigator — University Hospital, Bordeaux; Michel GUINOT, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Prétagut, CHU Nantes, France